CLINICAL TRIAL: NCT03448133
Title: Repetitive Transcranial Magnetic Stimulation for the Treatment of Primary Progressive Aphasia: A Randomized Controlled Tria
Brief Title: rTMS for the Treatment of Primary Progressive Aphasia: A Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the expiration of the previous ethical approval documents
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMSPPA-PUMCH
Record Dates: First submitted 2018-02-10; First posted 2018-02-27 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Aphasia, Primary Progressive; Repetitive Transcranical Magnetic Stimulation
MeSH Terms: conditions — Aphasia, Primary Progressive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS treatment group (Experimental): The participants will be devided into rTMS treatment and sham treatment by means of randomized methods.The protocol of treatment is to use rTMS with high frequency 10/20Hz 120%RMT 20 times for one month. The device is Magtism rTMS made in London, UK
  Interventions: Device: Magstim rTMS
- sham treatment group (Sham Comparator): The control group is to receive sham treatment. The device is the same as the one used in the real treatment group.
  Interventions: Device: Magstim rTMS

INTERVENTIONS:
Device: Magstim rTMS — The device is made in London,UK

SUMMARY:
The primary progressive aphasia (PPA) is a neurodegenerative condition characterized by a gradual, irreversible decline of language function (Mesulam, 2001). There are no known treatments for PPA so far. The relentless progression of PPA symptoms eventually leads to a profound impairment in communication ability and, ultimately, to more generalized deficits of cognition. Some cases and small studies reported that Transcranial Magnetic Stimulation (TMS), one of the non-invasive neuromodulation tech, can be employed to facilitate language production and improve the language ability in patients with PPA. Herein we will explore the tolerance and efficacy of TMS for the treatment of PPA by the randomized controlled trial .Meanwhile the functional MRI tech will be used to investigate the neural network changing in the procedure

ELIGIBILITY:
Inclusion Criteria:

All participants had also been evaluated previously by a behavioral neurologist at the Peking Union Medical College Hospital and had been clinically diagnosed with a variant of PPA.

Exclusion Criteria:

1. Scored below 15 on the mini-mental state exam (MMSE) due to concerns that global cognitive impairment might preclude their ability to follow the directions and interfere with task performance.
2. Had a history of seizures or unexplained loss of consciousness, pregnancy, surgical breach of the skull, or any other medical or surgical contraindication to receiving noninvasive brain stimulation.
3. Is unable to complete the treatment and evaluations

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Boston naming test evaluation | Baseline
  Assessment of the language production
Boston naming test evaluation | One month(just after 20 times rTMS treatment)
  Assessment of the language production
Western Aphasia Battery(WAB) Speech fluency | Baseline
  Assessment of the language production
Western Aphasia Battery(WAB) Speech fluency | One month(just after 20 times rTMS treatment)
  Assessment of the language production
Repetition Part of WAB | Baseline
  Assessment of the repetition ability
Repetition Part of WAB | One month(just after 20 times rTMS treatment)
  Assessment of the repetition ability
Word recognition Part of WAB | Baseline
  Assessment of the reading
Word recognition Part of WAB | One month(just after 20 times rTMS treatment)
  Assessment of the reading
Syntax comprehension Part of Bilingual Aphasia Battery( Standard modern Chinese version) | Baseline
  Assessment of the grammar ability
Syntax comprehension Part of Bilingual Aphasia Battery( Standard modern Chinese version) | One month(just after 20 times rTMS treatment)
  Assessment of the grammar ability

SECONDARY OUTCOMES:
fMRI parameters(strength, efficiency, clustering coefficient, and characteristic path length) | Baseline
  Graph theoretical analysis of the speech/language network
fMRI parameters(strength, efficiency, clustering coefficient, and characteristic path length) | One month(just after 20 times rTMS treatment)
  Graph theoretical analysis of the speech/language network